CLINICAL TRIAL: NCT02461992
Title: An Open-label, Single Dose Pharmacokinetic Study Of Xyntha (Moroctocog Alfa (Af-cc), Recombinant Factor Viii) In Male Chinese Subjects With Hemophilia A
Brief Title: Study of PF-05208756, Moroctocog Alfa (AF-CC), Xyntha For Male Chinese Subjects With Hemophilia A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Basic Science
Other Study IDs: B1831082; 2015-003685-88 (EudraCT Number)
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-07

CONDITIONS: Hemophilia A
Keywords: FVIII activity
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous infusion of Xyntha (Experimental): observation arm
  Interventions: Drug: Intravenous infusions of Xyntha

INTERVENTIONS:
Drug: Intravenous infusions of Xyntha — A single dose 50IU/kg dose of Xyntha administered by intravenous infusion within 10 minutes on Day 1

SUMMARY:
An open-label, single dose pharmacokinetic study of Xyntha (Moroctocog Alfa (AF-CC), Recombinant Factor VIII) in male Chinese subjects with hemophilia A

DETAILED DESCRIPTION:
The purpose of this study is to obtain pharmacokinetic profiles of FVIII:C after Xyntha administration in Chinese patients with severe hemophilia A, which is in support of the continued registration of Xyntha in China

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

1. Male Chinese subjects 6 years or older (weight >20 kg) with severe hemophilia A (factor VIII activity <1%) previously treated with > 150 exposure days to any FVIII-containing products.
2. Subjects should not have received an infusion of any FVIII products for at least 3 days (at least 72 hours) before the administration of Xyntha on Day 1.
3. Subjects must be in a non bleeding state before the administration of Xyntha on Day 1.
4. Evidence of a personally or legally acceptable representative (legally acceptable representative is only applicable to pediatric subjects) signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
5. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Current FVIII inhibitor or history of FVIII inhibitor (defined as > upper limit of normal (ULN) of the local reporting laboratory).
2. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or clinical findings at Screening.
3. Diagnosed with any other bleeding disorder in addition to hemophilia A.
4. Documented Human Immunodeficiency Virus (HIV).
5. Subjects anticipating elective surgery or other invasive procedure within 1 month following study entry.
6. Treatment with immunomodulatory therapy within 30 days or 5 half lives whichever is longer, prior to study entry or planned use for the duration of study participation.
7. Subjects with known hypersensitivity to the active substance or to any of the excipients of Xyntha.
8. Subjects with a known hypersensitivity to Chinese Hamster Ovary cell (CHO cell) proteins.
9. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat, if deemed necessary: significant hepatic or renal impairment (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 x ULN, or total bilirubin >2 x ULN or serum creatinine >2 x ULN), prothrombin time >1.5 x ULN, platelet count <80,000 L. Subjects with Gilbert's disease may be enrolled.
10. Unwilling or unable to follow the terms of the protocol.
11. Any condition which may compromise the subject's ability to comply with and/or perform study related activities or that poses a clinical contraindication to study participation, in the opinion of the investigator or sponsor.
12. A positive urine drug screen.
13. History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces (150 mL) of wine, 12 ounces (360 mL) of beer, or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
14. Treatment with an investigational drug within 30 days or 5 half lives preceding Day 1, whichever is longer.
15. Screening supine blood pressure 140 mm Hg (systolic) or 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If blood pressure (BP) is 140 mm Hg (systolic) or 90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
16. Screening supine 12 lead ECG demonstrating QTcF >450 or a QRS interval >120 msec msec. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTcF values should be used to determine the subject's eligibility.
17. Blood donation (excluding plasma donations) of approximately 500 mL or more within 56 days prior to dosing.
18. History of sensitivity to heparin or heparin induced thrombocytopenia.
19. Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
20. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.
21. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
22. Subjects with history of infection within 1 week prior to study entry.
23. Male subjects with partners currently pregnant and male subjects able to father children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- China (2):
  - Phase I Unit, Clinical Pharmacology Research Center, Peking Union Medical College Hospital, Beijing
  - Hematology Department,Beijing Children's Hospital, Capital Medical University, Beijing

REFERENCES:
- [Derived] Liu H, Wu R, Hu P, Sun F, Xu L, Liang Y, Nepal S, Qu PR, Huard F, Korth-Bradley JM. An Open-label, Single-dose, Pharmacokinetic Study of Factor VIII Activity After Administration of Moroctocog Alfa (AF-CC) in Male Chinese Patients With Hemophilia A. Clin Ther. 2017 Jul;39(7):1313-1319. doi: 10.1016/j.clinthera.2017.05.344. Epub 2017 Jun 7. PMID 28601434
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1831082&StudyName=An%20Open-label%2C%20Single%20Dose%20Pharmacokinetic%20Study%20Of%20Xyntha%20%28moroctocog%20Alfa%20%28af-cc%29%2C%20Recombinant%20Factor%20Viii%29%20In%20Male%20Chinese%20Subjects%20With%20Hemophilia%20A

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited Chinese male participants that were age 6 years or older with severe hemophilia A (factor VIII [FVIII] activity <1%) previously treated with >150 exposure days to any FVIII-containing product.
Groups:
- Xyntha 50 IU/kg: Participants were administered a single dose of recombinant antihemophilic factor (Xyntha) at 50 international units per kilogram (IU/kg) infused intravenously over 10 minutes.
Period: Overall Study
Arm/Group | Xyntha 50 IU/kg
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants who received at least 1 dose of study drug.
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
Age, Customized [Number; unit: participants]
  6 to 11 years | 3 (19.6)
  12 to 17 years | 5
  18 to 44 years | 2
  45 to 64 years | 3
  Greater than or equal to 65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma FVIII Activity (Cmax)
Time Frame: Pre-dose and 0.25, 0.5, 1, 3, 6, 9, 24, 28, 32, 48, and 72 hours post-dose
Population: The pharmacokinetic (PK) parameter analysis population is defined as all participants enrolled and treated who have at least 1 of the PK parameters of primary interest reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/milliliter (mL)
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
IU/milliliter (mL) | 1.147 (44)

2. Primary Outcome: Area Under the Plasma FVIII Activity-Time Profile From Time 0 to Time of the Last Quantifiable Concentration (AUClast)
Time Frame: Pre-dose and 0.25, 0.5, 1, 3, 6, 9, 24, 28, 32, 48, and 72 hours post-dose
Population: The PK parameter analysis population is defined as all participants enrolled and treated who have at least 1 of the PK parameters of primary interest reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hour/mL
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
IU*hour/mL | 14.49 (57)

3. Primary Outcome: Area Under the Plasma FVIII Activity-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf)
Time Frame: Pre-dose and 0.25, 0.5, 1, 3, 6, 9, 24, 28, 32, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hour/mL
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
IU*hour/mL | 15.21 (58)

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Pre-dose and 0.25, 0.5, 1, 3, 6, 9, 24, 28, 32, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
hour | 0.500 [0.250 to 3.00]

5. Primary Outcome: Clearance (CL)
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pre-dose and 0.25, 0.5, 1, 3, 6, 9, 24, 28, 32, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hour/kg
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
mL/hour/kg | 3.295 (56)

6. Primary Outcome: Volume of Distribution at Steady-State (Vss)
Description: Volume of distribution is the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss is the volume of distribution at steady-state.
Time Frame: Pre-dose and 0.25, 0.5, 1, 3, 6, 9, 24, 28, 32, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
mL/kg | 53.96 (29)

7. Primary Outcome: Terminal Phase Rate Constant (Kel)
Description: Terminal phase rate constant is the absolute value of the slope of a linear regression during the terminal phase of the natural--logarithm transformed concentration--time profile.
Time Frame: Pre-dose and 0.25, 0.5, 1, 3, 6, 9, 24, 28, 32, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
1/hour | 0.06039 (39)

8. Primary Outcome: Terminal Elimination Half-Life (t1/2)
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose and 0.25, 0.5, 1, 3, 6, 9, 24, 28, 32, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
hour | 12.24 (4.4172)

9. Primary Outcome: Mean Residence Time (MRT)
Description: MRT = AUMCinf / AUCinf, where AUMCinf is the area under the first moment curve from zero time to infinity calculated as AUMCinf = AUMCt + ((t x Ct) / kel) + (Ct / kel^2). AUMCt is the area under the first moment curve from zero time to time t calculated using the trapezoidal method.
Time Frame: Pre-dose and 0.25, 0.5, 1, 3, 6, 9, 24, 28, 32, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
hour | 16.37 (38)

10. Primary Outcome: Incremental Recovery (INCREC)
Description: Incremental recovery is the increase in circulating FVIII activity for every IU of Xyntha administered per kilogram of body weight.
Time Frame: Pre-dose and 0.25, 0.5, 1, 3, 6, 9, 24, 28, 32, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/deciliter (dL) per IU/kg
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
IU/deciliter (dL) per IU/kg | 2.284 (44)

11. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to Day 28
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
participants
  Number of participants with AEs | 4 (44)
  Number of participants with SAEs | 2

12. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities Meeting the Criteria for Potential Clinical Concern
Description: The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell count, RBC morphology, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, and total protein; urinalysis (pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy [if urine dipstick was positive for blood, protein, nitrites or leukocyte esterase]); others (urine drug screening, FVIII inhibitor assay, FVIII activity, prothrombin time [PT], activated partial thromboplastin time [APTT], anti-human immunodeficiency virus [HIV] 1, hepatitis C virus antibody [HCVAb], HAVAb, HBsAg, HBsAb, HBcAb). Only parameters which met abnormality criteria are reported.
Time Frame: Baseline up to Day 4
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
participants
  APTT >1.1X upper limit of normal (ULN) | 13 (44)
  Potassium <0.9X lower limit of normal (LLN) | 1
  Urine leukocyte >=1 | 1

13. Other Pre Specified Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Findings
Description: Vital signs assessment included pulse rate and blood pressure. Criteria for vital sign values meeting potential clinical concern included: supine pulse rate <50 beats per minute (bpm), >=30 bpm increase from baseline, or >25 bpm decrease from baseline; systolic blood pressure (SBP) <90 milliliters of mercury (mmHg), >=30 mmHg increase from baseline, or >=30 mmHg decrease from baseline; diastolic blood pressure (DBP) <50 mmHg, >=20 mmHg increase from baseline, or >=20 mmHg decrease from baseline.
Time Frame: Baseline up to Day 4
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
participants
  Supine SBP <90 mmHg | 0 (44)
  Supine DBP <50 mmHg | 0
  Supine Pulse Rate <50 bpm | 0
  Supine SBP >=30 mmHg Increase From Baseline | 0
  Supine DBP >=20 mmHg Increase From Baseline | 0
  Supine Pulse Rate >=30 bpm Increase From Baseline | 1
  Supine SBP >=30 mmHg Decrease From Baseline | 0
  Supine DBP >=20 mmHg Decrease From Baseline | 0
  Supine Pulse Rate >=25 bpm Increase From Baseline | 0

14. Other Pre Specified Outcome: Number of Participants With Positive FVIII Inhibitor Activity at Day 4
Description: As with all FVIII products, participants using Xyntha were monitored for the development of FVIII inhibitors. Values >= 0.6 Bethesda Unit (BU) per mL were considered positive results.
Time Frame: Day 4
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Xyntha 50 IU/kg
Number analyzed (Participants) | 13
participants | 2 (44)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 28
Arm/Group | Xyntha 50 IU/kg
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xyntha 50 IU/kg (N=13)
Factor VIII inhibition (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xyntha 50 IU/kg (N=13)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.